CLINICAL TRIAL: NCT04281420
Title: A Phase I Open-Label Study of the Safety and Tolerability of ATG-019, a Dual Inhibitor of PAK4 and NAMPT, in Patients With Advanced Solid Tumors or Non-Hodgkin's Lymphoma
Brief Title: A Study of Evaluating Dual Inhibitor of PAK4 and NAMPT ATG-019 in Advanced Solid Tumors or Non-Hodgkin's Lymphoma
Acronym: TEACH
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Because the sponsor modified the study-product development strategy.
Sponsor: Antengene Therapeutics Limited (Industry)
Responsible Party: Sponsor
Organization: Antengene Corporation (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATG-019-STL-001
Record Dates: First submitted 2020-02-18; First posted 2020-02-24 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2022-07

CONDITIONS: Solid Tumor, Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — KPT-9274

STUDY DESIGN:
Intervention Model Description: ATG-019 ATG-019+Niacin ER
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATG-019 Alone (Experimental): A starting does of 30 mg QoD×3 ATG-019
  Interventions: Drug: ATG-019
- ATG-019 + Niacin ER (Experimental): A starting dose of 60 mg ATG-019 and 500 mg niacin ER
  Interventions: Combination Product: ATG-019 + Niacin ER

INTERVENTIONS:
Drug: ATG-019 — ATG-019 30 mg QoD×3 is selected as the staring dose. Oral ATG-019 will be taken three times a week every other day (Days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26) during each 28-day cycle.
  Other Names: KPT-9274
  Arms: ATG-019 Alone
Combination Product: ATG-019 + Niacin ER — ATG-019 60 mg is selected as starting dose. Oral ATG-019 will be taken three times a week every other day (Days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26) during each 28-day cycle. And a starting dose of 500 mg niacin ER (may be titrated up to 1,000 mg of daily dose, per label) co-administered with each dose of ATG-019.
  Arms: ATG-019 + Niacin ER

SUMMARY:
This is a multi-center, open-label clinical study with separate Dose Escalation and Expansion Phases to assess preliminary safety, tolerability, and efficacy of ATG-019, a dual inhibitor of PAK4 and NAMPT, alone or co-administered with starting dose of 500 mg niacin ER in patients with advanced solid tumors or non-Hodgkin's lymphoma (NHL).

DETAILED DESCRIPTION:
This is a multi-center, open-label clinical study with separate Dose Escalation and Expansion Phases to assess preliminary safety, tolerability, and efficacy of ATG-019, a dual inhibitor of PAK4 and NAMPT, alone or co-administered with starting dose of 500 mg niacin ER (may be titrated to 1,000 mg of daily dose, per label), in patients with advanced solid tumors or non-Hodgkin's lymphoma (NHL) for which all standard therapeutic options considered useful by the investigator have been exhausted and with PD at study entry. The MTD and RP2D will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any screening procedures and in accordance with local and institutional guidelines.
2. Age ≥18 years.
3. Patients with histologically or cytologically confirmed, NHL or advanced solid tumors which have progressed despite standard therapy, for whom no standard therapy exists, or who have refused standard therapy.
4. Patients must have objective evidence of PD on study entry:

   1. Advanced solid tumors: Measureable disease as defined by RECIST 1.11.
   2. NHL: Measureable disease including target lesion(s) as defined by the Cheson 2014 Classification2 for initial evaluation and staging.
5. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
6. Adequate hepatic function.
7. Adequate renal function.
8. Life expectancy of ≥ 3 months.
9. Adequate hematopoietic function.
10. Female patients of child-bearing potential must agree to use dual methods of contraception (including one highly effective and one effective method of contraception) and have a negative serum pregnancy test at Screening, and male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential.

Exclusion Criteria:

1. Female patients who are pregnant or lactating.
2. Time since the last prior therapy for treatment of advanced solid tumors or NHL**:

   1. Radiation, chemotherapy, immunotherapy or any other anticancer therapy, including investigational anti-cancer therapy ≤ 4 weeks prior to C1D1.
   2. Palliative steroids for disease related symptoms within 7 days prior to C1D1.
3. Known central nervous system metastases.
4. Major surgery within 4 weeks before C1D1.
5. Impaired cardiac function or clinically significant cardiac diseases.
6. Active infection with completion of therapeutic antibiotics, antivirals, or antifungals within 1 week prior to C1D1.
7. Patients diagnosed with tuberculosis and had received treatment.
8. Patients with a known history of human immunodeficiency virus (HIV).
9. Known, active hepatitis A, B, or C infection.
10. Serious psychiatric or medical conditions that, in the opinion of the Investigator, could interfere with treatment, compliance, or the ability to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
To determine MTD* or RP2D* | 18 months
  MTD will be evaluated using the NCI-CTCAE, Version 5.0; RP2D will be determined by SMC for dose escalation phase.
To evaluate the Dose-Limiting Toxicity (DLT) for dose escalation phase | 18 months
  DLTs will be evaluated using the CTCAE, Version 5.0 for grading.
Overall Response Rate (ORR) | 18 months
  ORR analysis will be performed for both study phases by calculating the point estimate of the percentage of patients who have either CR or PR, presented as the number and percentage of patients, including a two-sided 95% CI.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 18 months
  To determine the maximum plasma concentration (Cmax) for dose escalation phase.
Time to Reach Cmax （Tmax） | 18 months
  To evaluate the time to reach Cmax after single and multiple doses for dose escalation phase.
To determine RP2D* | 18 months
  RP2D will be determined by SMC for dose escalation phase.
Duration of response (DOR) | 18 months
  The duration of time from first meeting CR or PR measurement criteria (whichever occurs first) until the first date that PD recurrence is objectively documented.
Disease control rate (DCR) | 18 months
  The analysis of DCR will be similar to that described for ORR, for patients who achieve CR, PR, or SD for ≥ 8 weeks.
Progression-free survival (PFS) | 18 months
  The duration of time from date of first dose of study treatment until the first date that PD is objectively documented or death due to any cause.
Overall Survival (OS) | 18 months
  The duration of time from date of first dose of study treatment until death from any cause.
Time to progression (TTP) | 18 months
  The duration of time from date of first dose of study treatment to date of PD.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Xie, MD; PhD, Study Director — Medical Monitor
Locations (8):
- China (3):
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Fudan University Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated To Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital (KMUH), Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital (CGMHKS), Kaohsiung City
  - China Medical University Hospital (CMUH), Taichang
  - National Cheng Kung University Hospital (NCKUH), Tainan
  - Tri-Service General Hospital (TSGH), Taipei